CLINICAL TRIAL: NCT01159483
Title: A Phase I, First-in-Human, Randomized, Subject and Investigator-Blind, Sponsor Open, Single Escalating Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Pf-04958242 in Healthy Adult Volunteers
Brief Title: First-in-Human Study of PF-04958242 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B1701001
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Period 1: Participants received 0.01 milligrams (mg) of PF-04958242 or matching placebo, once, orally.
  Period 2: Participants received 0.03 mg of PF-04958242 or matching placebo, once, orally.
  Period 3: Participants received 0.1 mg of PF-04958242 or matching placebo, once, orally.
  Interventions: Drug: PF-04958242; Drug: Placebo
- Cohort B (Experimental): Period 1: Participants received 0.3 mg of PF-04958242 or matching placebo, once, orally (fasted).
  Period 2: Participants received 0.6 mg of PF-04958242 or matching placebo, once, orally.
  Period 3: Participants received 1.0 mg of PF-04958242 or matching placebo, once, orally (fed).
  Interventions: Drug: PF-04958242; Drug: Placebo

INTERVENTIONS:
Drug: PF-04958242 — Administered as specified in the treatment arm
Drug: Placebo — Administered as specified in the treatment arm

SUMMARY:
The primary objective of this study will evaluate the safety and tolerability of single, escalating doses of PF-04958242 administered orally to healthy adult participants. This study will also evaluate the plasma pharmacokinetics (PK) of single doses of PF-04958242 after single escalating doses of PF-04958242 administered orally to healthy adult participants.

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kilograms per meter quared (kg/m2);
* Total body weight >50 kilograms (kg) (110 pounds [lbs]);

Key Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing);
* Positive urine drug screen;
* Pregnant or nursing females, and females of child bearing potential;
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07-15 (Actual); Primary Completion 2010-10-16 (Actual); Study Completion 2010-10-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Baseline to Day 4
  An adverse event is any untoward medical occurrence in a clinical investigation subject administered a product or medical device. A serious adverse event or serious adverse drug reaction is any untoward medical occurrence at any dose that: Results in death; Is life-threatening (immediate risk of death); Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability/incapacity; Results in congenital anomaly/birth defect.
Maximum Observed Plasma Concentration (Cmax) | Day 1 and at multiple time points up to Day 4
Time to Reach Cmax (Tmax) | Day 1 and at multiple time points up to Day 4
Area Under the Concentration-Time Curve from Time 0 Extrapolated to Infinity (AUC0-inf) | Day 1 and at multiple time points up to Day 4
Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) | Day 1 and at multiple time points up to Day 4
Apparent Total Plasma Clearance (CL/F) | Day 1 and at multiple time points up to Day 4
Apparent Terminal Elimination Half-life (t½) | Day 1 and at multiple time points up to Day 4
Area Under the Plasma Drug Concentration-Time Curve up to the Last Quantifiable Time-Point (AUC0-last) | Day 1 and at multiple time points up to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Singapore, Singapore